CLINICAL TRIAL: NCT00166322
Title: Dopaminergic Neurotransmission in Schizophrenia, Patients at Risk and Healthy Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ludwig-Maximilians - University of Munich (Other)
Responsible Party: O. Pogarell, MD, University of Munich
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: DYN-SPECT-Pogarell; EK076/03
Record Dates: First submitted 2005-09-09; First posted 2005-09-14 (Estimated); Last update posted 2008-05-07 (Estimated); Status verified 2008-05

CONDITIONS: Schizophrenia
Keywords: IBZM-SPECT; Amphetamine Challenge; Schizophrenia; dopaminergic neurotransmission; Persons at risk for the development of schizophrenia; healthy subjects
MeSH Terms: conditions — Schizophrenia

INTERVENTIONS:
Procedure: IBZM-SPECT (bolus and constant infusion paradigm) — single IBZM-SPECT assessment at study inclusion

SUMMARY:
This study is an investigation of the dopaminergic neurotransmission in patients with schizophrenia, patients at risk for the development of schizophrenia, and healthy controls using an iodobenzamide-single photon emission computed tomography (IBZM-SPECT) imaging technique under amphetamine challenge.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of schizophrenia (currently unmedicated)
* Subjects at risk for the development of schizophrenia (prodromal symptoms)
* Healthy subjects
* Written informed consent

Exclusion Criteria:

* Neurological or severe somatic disorders
* Women during pregnancy or lactation
* Occupational exposition to radiation > 15mSv
* Medication known to interfere with IBZM
* Contraindications for the use of amphetamine challenge

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2004-01; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
dopamine receptor availability | cross-sectional

CONTACTS AND LOCATIONS:
Overall Officials: Oliver Pogarell, MD, Principal Investigator — Dept. of Psychiatry, University of Munich; Klaus Tatsch, MD, Principal Investigator — Dept. of Nuclear Medicine, University of Munich
Locations (2):
- Germany (2):
  - Dept. of Psychiatry, Munich
  - Dept. of Nuclear Medicine, Munich